CLINICAL TRIAL: NCT06890624
Title: Chinese Modified FOLFOXIRI Combined with PD-1 Inhibitor Versus MFOLFOX6 As Neoadjuvant Therapy for Locally Advanced Colon Cancer (cT4/N2): a Multicenter, Randomized, Controlled, Phase II Trial
Brief Title: MFOLFOXIRI Plus PD-1 Inhibitor Vs MFOLFOX6 As Neoadjuvant Therapy for Locally Advanced Colon Cancer
Acronym: OPTICAL-3
Status: Not yet recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Sun Yat-sen University (Other)
Responsible Party: Principal Investigator, Yanhong Deng, Professor, Sixth Affiliated Hospital, Sun Yat-sen University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: CSWOG-C06; C06 (Other: CSWOG)
Record Dates: First submitted 2025-03-17; First posted 2025-03-24 (Actual); Last update posted 2025-03-27 (Actual); Status verified 2025-03

CONDITIONS: Colon Cancer (stage II & III)
Keywords: colon cancer
MeSH Terms: conditions — Colonic Neoplasms | interventions — Immune Checkpoint Inhibitors

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- cmFOLFOXIRI plus PD-1 inhibitor (Experimental): cmFOLFOXIRI: oxaliplatin 85 mg/m² , irinotecan 150 mg/m², folinic acid 400 mg/m², 5-FU 2400 mg/m² continuous 46h infusion, repeat once every 2 weeks. PD-1 inhibitor 200mg, repeat once every 2 weeks. For 4 cycles before surgery.
  Interventions: Drug: cmFOLFOXIRI plus PD-1 inhibitor
- mFOLFOX6 (Active Comparator): mFOLFOX6: oxaliplatin 85 mg/m2, leucovorin 400 mg/m2, 5-FU 400 mg/m2 IV bolus, followed by 2400 mg/m2 continuous IV infusion over 46 hours, repeat once every 2 weeks. For 4 cycles before surgery.
  Interventions: Drug: mFOLFOX6

INTERVENTIONS:
Drug: cmFOLFOXIRI plus PD-1 inhibitor — cmFOLFOXIRI: oxaliplatin 85 mg/m² , irinotecan 150 mg/m², folinic acid 400 mg/m², 5-FU 2400 mg/m² continuous 46h infusion, repeat once every 2 weeks. PD-1 inhibitor 200mg, repeat once every 2 weeks.
  Arms: cmFOLFOXIRI plus PD-1 inhibitor
Drug: mFOLFOX6 — mFOLFOX6: oxaliplatin 85 mg/m2, leucovorin 400 mg/m2, 5-FU 400 mg/m2 IV bolus, followed by 2400 mg/m2 continuous IV infusion over 46 hours, repeat once every 2 weeks.
  Arms: mFOLFOX6

SUMMARY:
In patients with high-risk stage II and stage III colon cancer, curative surgery followed by adjuvant chemotherapy with FOLFOX or CAPOX regimens has become the standard treatment. However, 20 to 30% of these patients will develop distant metastasis, which ultimately results in death. In contrast to rectal cancer, the role of preoperative therapy in colon cancer is less well established. Relatively few phase III trials of preoperative therapy have been reported, although current NCCN guidelines do recommend neoadjuvant chemotherapy with FOLFOX or CAPOX regimen as an option for bulky T4b tumors. Neoadjuvant chemotherapy is an attractive approach for several reasons. The ability to deliver systemic therapies earlier in the treatment course to eradicate micrometastatic disease is conceptually appealing. In addition, surgery can stimulate tumor proliferation through inflammation and other immune pathways. Preoperative delivery of chemotherapy may also lead to higher rates of R0 resections, and chemotherapy tolerance can be better in the neoadjuvant setting, especially in colorectal surgeries that require prolonged recovery.

In the phase III study of the FOxTROT trial, the pCR rate for 6 weeks of neoadjuvant FOLFOX chemotherapy was only 4%, and a moderate or greater tumor regression was reported in 21% of patients in the NAC group. Our team also conducted the phase III OPTICAL trial, which utilized a longer period of NAC (12 weeks) with FOLFOX or CAPOX. In this trial, the pCR rate for the neoadjuvant chemotherapy group was 7%, and the downstaging rate (ypT0-2N0) was 20%. However, for patients with locally advanced colon cancer, particularly those with T4b and bulky nodal disease, the use of oxaliplatin- and fluoropyrimidine-based doublet chemotherapy does not adequately meet the clinical need for tumor shrinkage and downstaging. There is an urgent need to explore drugs with different mechanisms of action in combination with chemotherapy to improve efficacy.

DETAILED DESCRIPTION:
This trial is a two-arm, multicenter, open-label, prospective, randomized phase II study. Eligible patients with locally advanced (T4 or N2) colon cancer will be randomly assigned in a 1:1 ratio to receive either cmFOLFOXIRI plus a PD-1 inhibitor or mFOLFOX6 as neoadjuvant treatment.

ELIGIBILITY:
Inclusion Criteria:

1. Willing and able to provide written informed consent.
2. Histological or cytological documentation of adenocarcinoma of the colon (≥ 12 cm from the anal verge).
3. Determined preoperatively by either spiral or multidetector CT: T4 or N2.
4. Male or female subjects > 18 years < 70 of age.
5. Eastern Cooperative Oncology Group (ECOG) performance status of 0 or 1.
6. CT or MRI scans (done within 30 days of registration) of the chest, abdomen and pelvis all without clear evidence of distant metastatic (M1) disease.
7. No clinically significant obstruction, perforation, or bleeding related to the primary tumor.
8. No previous any systemic anticancer therapy for colon cancer disease.
9. Adequate bone marrow, hepatic and renal function as assessed by the following laboratory requirements conducted within 7 days of starting study treatment

Exclusion Criteria:

1. Previous or concurrent cancer that is distinct in primary site or histology from colon cancer within 5 years prior to randomization.
2. Significant cardiovascular disease including unstable angina or myocardial infarction within 6 months before initiating study treatment.
3. Heart failure grade III/IV (NYHA-classification).
4. Unresolved toxicity higher than CTCAE v.5.0 Grade 1 attributed to any prior therapy/procedure.
5. Subjects with known allergy to the study drugs or to any of its excipients.
6. Current or recent (within 4 weeks prior to starting study treatment) treatment of another investigational drug or participation in another investigational study.
7. Breast- feeding or pregnant women
8. Lack of effective contraception.

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 138 (Estimated)
Dates: Start 2025-05-01 (Estimated); Primary Completion 2027-05-01 (Estimated); Study Completion 2030-05-01 (Estimated)

PRIMARY OUTCOMES:
Pathologic complete response rate | 1 year
  The percentage of subjects with no residual viable tumor in the resected primary tumor specimen and all sampled regional lymph nodes after radical surgery (ypT0N0).

SECONDARY OUTCOMES:
R0 resection rate | 1 year
  The proportion of patients whose tumors are completely removed without residual cancer cells under the microscope. None of the following conditions can be considered as R0 resection: non-complete resection of the tumor, positive circumferential, proximal, or distal resection margin (resection margin of >1 mm).
Event-free survival (EFS) | 3 years
  The time between randomization and one of the following events: locally progressive disease leading to an unresectable tumor, local R2 resection, local recurrence after an R0/1 resection, distant metastases, a new primary colorectal cancer, or death from any cause, whichever occurred first.
Disease-free survival (DFS) | 3 years
  The time from the date of surgery to the date of locoregional recurrence, distant metastases, a new primary colorectal cancer, or death from any cause, whichever occurred first.
Overall survival (OS) | 5 years
  The time from randomization to death from any cause. Subjects who are still alive at the time of the analysis will be censored for OS on the latest known survival date.

IPD SHARING:
Plan to Share IPD: No